CLINICAL TRIAL: NCT02622334
Title: A MULTIPLE-CENTER, INVESTIGATOR/SUBJECT MASKED, ADAPTIVE, MULTIPLE ASCENDING DOSE, RANDOMIZED, PLACEBO-CONTROLLED, PARALLEL STUDY TO INVESTIGATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF RO5093151 FOLLOWING 7 DAYS ADMINISTRATION IN PATIENTS WITH PRIMARY OPEN ANGLE GLAUCOMA OR OCULAR HYPERTENSION
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO5093151 in Patients With Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP30002
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Part A (Experimental): Participants will receive up to 3 multiple ascending dose levels with the starting dose of 0.1% RO5093151 (topical ocular instillation) and sequentially 0.5% and 1% RO5093151 doses or placebo (3:1, active:placebo) twice a day (BID) on Day 1 and once a day (QD) for 6 days.
  Interventions: Drug: Placebo; Drug: RO5093151
- Part B (Experimental): Participants will receive highest feasible dose (HFD) or maximum tolerated dose (MTD) of RO5093151 from Part A or 0.005% latanoprost (topical ocular instillation) once daily for 7 days.
  Interventions: Drug: Latanoprost; Drug: RO5093151

INTERVENTIONS:
Drug: Latanoprost — Latanoprost is a ophthalmic solution, available in dose strength as 0.005%.
  Arms: Part B
Drug: Placebo — Matching placebo formulation will be administered in Part A.
  Arms: Part A
Drug: RO5093151 — RO5093151 is a ophthalmic solution, available in dose strengths as 0.1%, 0.5% and 1%.

SUMMARY:
The purpose of the study is to assess the safety, tolerability, and IOP effects of RO5093151 following 7 days of topical ocular treatment in patients with primary open angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ocular hypertension (OHT) or primary open angle glaucoma (POAG) in at least one eye (qualifying eye) as determined by the Investigator at screening or based on a reliable and documented assessment done within the last 6 months prior to screening provided that no progression of visual field damage is expected
* At baseline visit, intraocular pressure (IOP) >= 24 mmHg in the morning and >= 21 mmHg in the afternoon measurement in at least one eye (qualifying eye = study eye) and =< 34 mmHg at all time points in both eyes
* Best corrected logMAR visual acuity score of 0.7 (20/100 Snellen) or better in each eye as measured by ETDRS visual acuity test at screening
* Central corneal pachymetry measurement 420 to 620 micrometer in qualifying eye at screening
* Cup-to-disk ratio =< 0.8 (both eyes) at screening
* Anterior chamber angle is open and non-occludable as confirmed by the Investigator by gonioscopy examination at screening

Exclusion Criteria:

* History of any clinically significant gastrointestinal, renal, hepatic, bronchopulmonary, neurological, psychiatric, cardio-vascular, endocrinological, hematological or allergic disease (multiple allergies, seasonal allergy is acceptable), metabolic disorder, cancer or cirrhosis
* Uncontrolled hypertension (SBP >= 160 mmHg and/or DBP >= 100 mmHg) despite treatment at the time of screening confirmed by the average of >= 3 blood pressure measurements, properly measured with well-maintained equipment
* Clinically significant abnormalities in laboratory test results at screening
* Hypersensitivity to RO5093151 or any of the components of its formulation, or hypersensitivity to latanoprost or any of the components of its formulation (Part B only)
* Donation of blood over 500 mL within three months prior to screening
* Positive result on hepatitis B (HBV), hepatitis C (HCV), or HIV 1 and 2
* Presence of narrow angle (=< grade 2 Shaffer gonioscopic classification) or complete or partial closure, as measured by gonioscopy or at risk for angle closure as assessed by the Investigator
* Other forms of glaucoma than POAG or OHT in the study eye
* Any abnormality preventing reliable applanation tonometry
* Any clinically significant corneal scarring, haze or opacity
* Patient uncooperativeness that restricts adequate examination of IOP, ocular fundus or anterior chamber
* Evidence of clinically significant blepharitis, concurrent infectious/non-infectious conjunctivitis, keratitis or uveitis
* History or signs of penetrating ocular trauma. Uneventful (uncomplicated) cataract surgery performed 3 months prior to screening is allowed
* According to the Investigator's best judgment, risk of visual field or visual acuity worsening in either eye as a consequence of glaucoma progression or consequence of participation in the trial (i.e., during washout of ocular hypotensive medications or treatment with placebo) or any other ocular disease
* Unable to safely stop ocular hypotension medications prior to randomization according to the required minimum washout periods
* History of any ocular filtering surgical intervention, previous glaucoma intraocular surgery, or laser trabeculoplasty
* History of refractive surgery (laser assisted in-situ keratomileusis, laser epithelial keratomileusis, photorefractive keratectomy, phototherapeutic keratectomy)
* Any other intraocular surgery within 6 months of screening
* Advanced age-related macular degeneration (wet or dry), vitreous hemorrhage, diabetic retinopathy or any progressive retinal or optic nerve disease from any cause other than glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 12 weeks
Changes in vital signs, electrocardiogram (ECG), opthalmologic assessments, and clinical laboratory results | Up to 12 weeks
Change in mean IOP after 7 days treatment vs baseline: change from baseline for RO5093151 and latanoprost and difference in change from baseline between RO5093151 and latanoprost | Baseline (Day 1) and Day 8

SECONDARY OUTCOMES:
Change in IOP at matched clock-times after 7 days of treatment vs baseline (diurnal IOP) and between RO5093151 and latanoprost | Baseline and Day 8
Maximum observed plasma concentration (Cmax) | Day 1: Pre-dose (morning); 30 minutes, 1, 4, 8, 11 (evening pre-dose) and 12 hours post-dose; Day 7: Pre-dose (evening), 1, 12 (Day 8), 16 (Day 8), 20 (Day 8) hours post-dose
Time to maximum observed plasma concentration (Tmax) | Day 1: Pre-dose (morning); 30 minutes, 1, 4, 8, 11 (evening pre-dose) and 12 hours post-dose; Day 7: Pre-dose (evening), 1, 12 (Day 8), 16 (Day 8), 20 (Day 8) hours post-dose
Concentration at the end of a dosing interval before the next dose administration (Ctrough) | Day 1: Pre-dose (morning); 30 minutes, 1, 4, 8, 11 (evening pre-dose) and 12 hours post-dose; Day 7: Pre-dose (evening), 1, 12 (Day 8), 16 (Day 8), 20 (Day 8) hours post-dose
Area under the plasma concentration versus time curve from zero to 24 h post-dose (AUC0-24) | Day 1: Pre-dose (morning); 30 minutes, 1, 4, 8, 11 (evening pre-dose) and 12 hours post-dose; Day 7: Pre-dose (evening), 1, 12 (Day 8), 16 (Day 8), 20 (Day 8) hours post-dose
Area under the plasma concentration versus time curve up to the last measurable concentration (AUClast) | Day 1: Pre-dose (morning); 30 minutes, 1, 4, 8, 11 (evening pre-dose) and 12 hours post-dose; Day 7: Pre-dose (evening), 1, 12 (Day 8), 16 (Day 8), 20 (Day 8) hours post-dose
Apparent terminal half-life (T1/2) | Day 1: Pre-dose (morning); 30 minutes, 1, 4, 8, 11 (evening pre-dose) and 12 hours post-dose; Day 7: Pre-dose (evening), 1, 12 (Day 8), 16 (Day 8), 20 (Day 8) hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- United States (6):
  - Sall Research Medical Center, Artesia, California
  - Rocky Mountain Lions Eye Inst, Aurora, Colorado
  - Eye Care Centers Management, Inc. (Clayton Eye Center), Morrow, Georgia
  - New York Eye and Ear Infirmary of Mt. Sinai; New York Glaucoma Research Institute, New York, New York
  - Cornerstone Eye Care, Div of Cornerstone Health Care, High Point, North Carolina
  - West Virginia University Eye Institute, Morgantown, West Virginia
- Singapore National Eye Centre; Glaucoma Department, Singapore, Singapore